CLINICAL TRIAL: NCT00432133
Title: Behavioral 2X2 Randomized Controlled Trial to Determine Individual and Environmental Mechanisms of Physical Activity Behavior Change
Brief Title: Individual and Environmental Mechanisms of PA Change
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kaiser Permanente (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: DK70553; R01DK070553 (NIH); DK70553
Record Dates: First submitted 2007-02-05; First posted 2007-02-07 (Estimated); Last update posted 2012-04-27 (Estimated); Status verified 2012-04

CONDITIONS: Physical Activity; Behavior Change
Keywords: Physical Activity; Behavior Change; Mechanism; Environmental; Ecological Model of Physical Activity
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (Experimental): Protection motivation theory-based tailored intervention to promote physical activity delivered via interactive technology (computer interactive session, automated telephone counseling, tailored newsletters).
  Interventions: Behavioral: Protection Motivation Theory-Based Intervention
- 2 (Experimental): Environmental access and awareness intervention to promote physical activity delivered via interactive technology (computer interactive session, automated telephone counseling, tailored newsletters).
  Interventions: Behavioral: Environmenta
- 3 (Experimental): Combination intervention combining protection motivation and environmental intervention components to promote physical activity delivered via interactive technology (computer interactive session, automated telephone counseling, tailored newsletters).
  Interventions: Behavioral: Protection Motivation Theory-Based Intervention; Behavioral: Environmenta

INTERVENTIONS:
Behavioral: Protection Motivation Theory-Based Intervention — Targets perceptions of outcome severity and susceptibility, self-efficacy, response efficacy, response costs, and rewards of physical inactivity. One computer interactive session is followed by 3 automated telephone counseling sessions and 4 tailored newletters spread over a 6 month period.
  Arms: 1; 3
Behavioral: Environmenta — Targets increased awareness and use of local parks and trials near the home and work environments. Targets increased access by providing membership to a local fitness facility for 12 months. One computer interactive session is followed by 3 automated telephone counseling sessions and 4 tailored newletters spread over a 6 month period.
  Arms: 2; 3

SUMMARY:
The focus of this study is to determine the mechanisms that underlie Physical Activity behavior change. We have 2 primary objectives. One, to test the effectiveness of brief, practical interventions to promote and maintain Physical Activity among individuals who are referred to a treadmill stress test but do not present symptoms of cardiac disease. Two, to test the potential individual and environmental mediators and moderators of this effect.

DETAILED DESCRIPTION:
There is a dearth of information on the mechanisms, and potential moderators, of physical activity (PA) intervention effectiveness. Understanding the mechanisms of PA change will aid in successful intervention development while understanding moderators will allow a matching of intervention components to individual needs of particular populations. To definitively understand mechanisms and moderators of behavior change it is necessary to develop theory-based interventions that include specific strategies that target proposed mechanisms of change while monitoring the proposed mediating and moderating variables prior to and following intervention. This proposal highlights the use of the Ecological Model of Physical Activity (EMPA) as a theoretical guide to strategy development. The EMPA highlights the necessity to address individual (biological & psychosocial) and environmental variables (e.g., PA resource accessibility) when developing and implementing interventions. Health care patients who have been referred for a treadmill cardiovascular stress test-but do not present abnormal ECG or chest pain during testing-will be will be stratified by diagnosis of low heart rate recovery, a potential biological moderator of intervention effectiveness. To detect the potential independent and combined effects of individual motivation and environmental accessibility we will conduct a randomized 2X2 factorial trial to test proposed mediators of effectiveness. Participants (n=500) will be randomized to an individual (I), environmental (E) , combination (I+E), or matched contact nutrition control. All intervention conditions will include a CD-ROM session, 3 tailored mail, and 3 tailored automated telephone follow-ups over a 6-month period. We will assess the reach, effectiveness, clinician adoption, and staff implementation of these interventions, individually, in combination, and when compared to controls among an understudied and high need population-individuals who are at an elevated risk, but have not yet suffered a serious cardiac event (approximately 3,000,000 individuals/year in the US). The results of this project will identify the causal, and potentially additive, relationships of environmental and individual mediators of PA change and allow the examination of potential biological moderators of effectiveness. Because intervention typically effects decrease over time and studies do not address setting-related issues necessary to ensure sustainability of delivery at the organizational level we will determine the maintenance of intervention effects on causal mechanisms and PA, 6 & 12 months following intervention. The interventions will be developed for delivery within the regular scope of treadmill stress testing by typical medical staff and cost of delivery will be assessed for each intervention condition. This project uniquely utilizes methods that will facilitate institutionalization of the intervention components following the successful completion of the trial and potential adoption of the intervention in other health care settings.

ELIGIBILITY:
Inclusion Criteria:

* No chest pains during stress testing
* Normal ECG During Stress Testing.
* Inactive or insufficiently active (<150 moderate intensity PA/week)

Exclusion Criteria:

* Age
* No access to telephone
* Not able to read or understand English.
* Home and Work address outside of 6-county area
* Have an active recreation center membership
* Any other contraindication to physical activity identified during stress testing.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 452 (Actual)
Dates: Start 2006-02; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
Physical Activity: CHAMPS self report measure and Actigraph Accelerometers | 6 & 12 months

SECONDARY OUTCOMES:
Dollar amounts to include cost of intervention delivery by condition. | 6 months
Heart Rate Recovery. | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Paul A Estabrooks, PhD, Principal Investigator — Kaiser Permanente
Locations (1):
- Kaiser Permanente Colorado, Institute for Health Research, Denver, Colorado, United States

REFERENCES:
- [Derived] Almeida FA, Smith-Ray RL, Dzewaltowski DA, Glasgow RE, Lee RE, Thomas DS, Xu S, Estabrooks PA. An Interactive Computer Session to Initiate Physical Activity in Sedentary Cardiac Patients: Randomized Controlled Trial. J Med Internet Res. 2015 Aug 24;17(8):e206. doi: 10.2196/jmir.3759. PMID 26303347